CLINICAL TRIAL: NCT06435533
Title: Cold Atmospheric Plasma for the Endoscopic Treatment of Duodenal Polyps in Patients With Familial Adenomatous Polyposis
Acronym: coldAPC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Prof. Dr. Thomas Rösch, Prof. Dr. Thomas Roesch Medical Director, Interdisciplinary Endoscopy Department and Clinic University Hospital Hamburg-Eppendorf, Universitätsklinikum Hamburg-Eppendorf
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-101193-BO-ff
Record Dates: First submitted 2024-03-14; First posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Adenomatous Polyposis Coli; Familial Adenomatous Polyposis; Duodenal Adenoma
Keywords: Familial Adenomatous Polyposis; FAP; duodenal adenoma; argon plasma coagulation; Spigelman classification stage III
MeSH Terms: conditions — Adenomatous Polyposis Coli

STUDY DESIGN:
Intervention Model Description: peri-ampullary FAP polyps of size smaller than 10 mm will be treated with low energy argonplasma coagulation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- duodenal polyps <10 mm (Experimental): low energy argonplasma coagulation
  Interventions: Device: low energy argonplasma coagulation

INTERVENTIONS:
Device: low energy argonplasma coagulation — see above
  Other Names: cold APC

SUMMARY:
The objective of this study is to investigate the feasibility for the treatment of precancerous peri-ampullary FAP polyps in the duodenum using low-thermal argonplasma.

DETAILED DESCRIPTION:
Familial adenomatous polyposis (FAP) is an autosomal dominantly inherited disorder, which results from a germ line mutation in the APC (adenomatous polyposis coli) gene. FAP is characterized by the formation of very high number of colorectal adenomatous polyps which could cause the development of colorectal cancer in the 5th decade of life. After colon surgery patients are still at risk of developing upper GI cancer e.g. in the duodenum. Because of the continuing risk for the development of duodenal cancer, regular endoscopic surveillance is recommended for these patients.

In this study a new APC modality (Precise mode E1) applied for the remission of FAP polyps during routine endoscopic surveillance is suggested. Argonplasma coagulation (APC) is widely used for the ablation and coagulation of superficial lesions in the GI tract. The application of high thermal tissue destroying APC in the duodenum is challenging due to the anatomy of the duodenal wall which is thin and therefore susceptible to thermal damage.

The application of low-thermal argonplasma in the GI tract could be just as useful as it was suggested for the treatment of neoplastic tissue in gynecology. Low-thermal APC using Erbe Standard 3.2 mm FiAPC probe and Precise mode was successfully applied for the remission of cervical intraepithelial neoplasia. The formation of reactive oxygen and nitric oxide species has been discussed as trigger for the effect on neoplasia tissue of low-thermal argonplasma.

Regarding current knowledge this is the first application of this APC modality in the GI tract.

ELIGIBILITY:
Inclusion Criteria:

* confirmed FAP disease
* duodenal polyposis with recommendation of a follow-up EGD in 12 months corresponding to stage III (7-8 points) according to Spigelman
* presence of duodenal polyps < 10 mm
* written Informed Consent

Exclusion Criteria:

* presence of lesions that are suspicious of the presence of high-grade dysplasia or carcinoma
* pregnancy or breastfeeding
* severe general illnesses (permanent ASA (American Society of Anesthesiologists) III and IV) who do not prognostically benefit from follow-up, life expectancy < 1 year
* severe coagulopathy
* any visible state of duodenal surface that makes APC treatment impossible, e.g. inflammation, stricture, stenosis or scarring changes/scar areas

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-12-06 (Actual); Primary Completion 2025-01-30 (Estimated); Study Completion 2025-03-02 (Estimated)

PRIMARY OUTCOMES:
polyp number | 12 months
  Significant reduction in the number of duodenal polyps at the next follow-up appointment
polyp size | 12 months
  Significant reduction in the size of duodenal polyps at the next follow-up appointment

SECONDARY OUTCOMES:
acute haematemesis | 24 hours
  rate of acute adverse incidents: bleeding
acute hemoglobin drop | 24 hours
  rate of acute adverse incidents: Hb drop < 2g /dl (grammes per decilitre)
acute severe hemoglobin drop | 24 hours
  rate of acute adverse incidents: Hb drop = or > 2g /dl (grammes per decilitre)
blood transfusion | 24 hours
  rate of acute adverse incidents: Hb drop = or > 2g /dl (grammes per decilitre)
endoscopic hemostasis | 24 hours
  rate of acute adverse incidents: coagulation or clipping
treatment of perforation | 24 hours
  rate of acute adverse incidents: endoscopic clipping
need for surgical intervention | 24 hours
  rate of acute adverse incidents: bleeding or perforation which can not be handled by endoscopic treatment
acute abdominal pain | 24 hours
  rate of acute adverse incidents:pain
acute dysphagia | 24 hours
  rate of acute adverse incidents: stenosis
acute rise of temperature | 24 hours
  rate of acute adverse incidents: fever <38°C (degrees Centigrade)
EGD (esophago-gastro-duodenoscopy) time | during EGD; up to 45 minutes
  total EGD performing time
therapy time | up to 30 minutes
  total ablation time in minutes
abdominal pain | 4 days
  abdominal pain assessed by patient survey
nausea | 4 days
  nausea assessed by patient survey
feeling of fullness | 4 days
  feeling of fullness assessed by patient survey
emesis | 4 days
  emesis assessed by patient survey
signs of bleeding | 4 days
  hematemesis or tar faeces assessed by patient survey
fever | 4 days
  fever >38°C
need for physician help | 4 days
  visits in doctor's office or hospital
success rate | 12 months
  Change in stage/number of points in Spigelman classification compared to the previous examination
dysphagia | 12 months
  dysphagia caused by duodenal stricture
balloon dilatations | 12 months
  need for endoscopic dilatation of strictured duodenum
abdominal pain | 12 months
  general abdominal pain assessed by patient survey
postprandial pain | 12 months
  postprandial abdominal pain assessed by patient survey
emesis | 12 months
  regurgitation due to duodenal strictures assessed by EGD

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Rösch, Professor, Principal Investigator — Universitätskrankenhaus Hamburg-Eppendorf
Locations (1):
- University Hospital Hamburg-Eppendorf, Hamburg, Germany

REFERENCES:
- [Background] Aelvoet AS, Buttitta F, Ricciardiello L, Dekker E. Management of familial adenomatous polyposis and MUTYH-associated polyposis; new insights. Best Pract Res Clin Gastroenterol. 2022 Jun-Aug;58-59:101793. doi: 10.1016/j.bpg.2022.101793. Epub 2022 Mar 16. PMID 35988966
- [Background] Half E, Bercovich D, Rozen P. Familial adenomatous polyposis. Orphanet J Rare Dis. 2009 Oct 12;4:22. doi: 10.1186/1750-1172-4-22. PMID 19822006
- [Background] Ghorbanoghli Z, Bastiaansen BA, Langers AM, Nagengast FM, Poley JW, Hardwick JC, Koornstra JJ, Sanduleanu S, de Vos Tot Nederveen Cappel WH, Witteman BJ, Morreau H, Dekker E, Vasen HF. Extracolonic cancer risk in Dutch patients with APC (adenomatous polyposis coli)-associated polyposis. J Med Genet. 2018 Jan;55(1):11-14. doi: 10.1136/jmedgenet-2017-104545. Epub 2017 May 10. PMID 28490611
- [Background] Bulow S, Bjork J, Christensen IJ, Fausa O, Jarvinen H, Moesgaard F, Vasen HF; DAF Study Group. Duodenal adenomatosis in familial adenomatous polyposis. Gut. 2004 Mar;53(3):381-6. doi: 10.1136/gut.2003.027771. PMID 14960520
- [Background] Kadmon M, Tandara A, Herfarth C. Duodenal adenomatosis in familial adenomatous polyposis coli. A review of the literature and results from the Heidelberg Polyposis Register. Int J Colorectal Dis. 2001 Apr;16(2):63-75. doi: 10.1007/s003840100290. PMID 11355321
- [Background] Bjork J, Akerbrant H, Iselius L, Bergman A, Engwall Y, Wahlstrom J, Martinsson T, Nordling M, Hultcrantz R. Periampullary adenomas and adenocarcinomas in familial adenomatous polyposis: cumulative risks and APC gene mutations. Gastroenterology. 2001 Nov;121(5):1127-35. doi: 10.1053/gast.2001.28707. PMID 11677205
- [Background] van Leerdam ME, Roos VH, van Hooft JE, Dekker E, Jover R, Kaminski MF, Latchford A, Neumann H, Pellise M, Saurin JC, Tanis PJ, Wagner A, Balaguer F, Ricciardiello L. Endoscopic management of polyposis syndromes: European Society of Gastrointestinal Endoscopy (ESGE) Guideline. Endoscopy. 2019 Sep;51(9):877-895. doi: 10.1055/a-0965-0605. Epub 2019 Jul 23. PMID 31342472
- [Background] Spigelman AD, Williams CB, Talbot IC, Domizio P, Phillips RK. Upper gastrointestinal cancer in patients with familial adenomatous polyposis. Lancet. 1989 Sep 30;2(8666):783-5. doi: 10.1016/s0140-6736(89)90840-4. PMID 2571019
- [Background] Manner H. Thermal ablative therapies in the gastrointestinal tract. Curr Opin Gastroenterol. 2023 Sep 1;39(5):370-374. doi: 10.1097/MOG.0000000000000954. Epub 2023 Jun 22. PMID 37389449
- [Background] Manner H. Argon plasma coagulation therapy. Curr Opin Gastroenterol. 2008 Sep;24(5):612-6. doi: 10.1097/MOG.0b013e32830bf825. PMID 19122503
- [Background] Martusevich AK, Surovegina AV, Bocharin IV, Nazarov VV, Minenko IA, Artamonov MY. Cold Argon Athmospheric Plasma for Biomedicine: Biological Effects, Applications and Possibilities. Antioxidants (Basel). 2022 Jun 27;11(7):1262. doi: 10.3390/antiox11071262. PMID 35883753
- [Background] Marzi J, Stope MB, Henes M, Koch A, Wenzel T, Holl M, Layland SL, Neis F, Bosmuller H, Ruoff F, Templin M, Kramer B, Staebler A, Barz J, Carvajal Berrio DA, Enderle M, Loskill PM, Brucker SY, Schenke-Layland K, Weiss M. Noninvasive Physical Plasma as Innovative and Tissue-Preserving Therapy for Women Positive for Cervical Intraepithelial Neoplasia. Cancers (Basel). 2022 Apr 12;14(8):1933. doi: 10.3390/cancers14081933. PMID 35454839
- [Background] Grund KE, Storek D, Farin G. Endoscopic argon plasma coagulation (APC) first clinical experiences in flexible endoscopy. Endosc Surg Allied Technol. 1994 Feb;2(1):42-6. PMID 8081915
- [Background] Karamanolis G, Triantafyllou K, Tsiamoulos Z, Polymeros D, Kalli T, Misailidis N, Ladas SD. Argon plasma coagulation has a long-lasting therapeutic effect in patients with chronic radiation proctitis. Endoscopy. 2009 Jun;41(6):529-31. doi: 10.1055/s-0029-1214726. Epub 2009 May 13. PMID 19440956
- [Background] Peng M, Guo X, Yi F, Shao X, Wang L, Wu Y, Wang C, Zhu M, Bian O, Ibrahim M, Chawla S, Qi X. Endoscopic treatment for gastric antral vascular ectasia. Ther Adv Chronic Dis. 2021 Aug 12;12:20406223211039696. doi: 10.1177/20406223211039696. eCollection 2021. PMID 34408826
- [Background] Swanson E, Mahgoub A, MacDonald R, Shaukat A. Medical and endoscopic therapies for angiodysplasia and gastric antral vascular ectasia: a systematic review. Clin Gastroenterol Hepatol. 2014 Apr;12(4):571-82. doi: 10.1016/j.cgh.2013.08.038. Epub 2013 Sep 5. PMID 24013107
- [Background] Lienert A, Bagshaw PF. Treatment of duodenal adenomas with endoscopic argon plasma coagulation. ANZ J Surg. 2007 May;77(5):371-3. doi: 10.1111/j.1445-2197.2007.04063.x. PMID 17497979
- [Background] Manner H, May A, Faerber M, Rabenstein T, Ell C. Safety and efficacy of a new high power argon plasma coagulation system (hp-APC) in lesions of the upper gastrointestinal tract. Dig Liver Dis. 2006 Jul;38(7):471-8. doi: 10.1016/j.dld.2006.03.022. Epub 2006 May 15. PMID 16702032
- [Background] Jaganmohan S, Lynch PM, Raju RP, Ross WA, Lee JE, Raju GS, Bhutani MS, Fleming JB, Lee JH. Endoscopic management of duodenal adenomas in familial adenomatous polyposis--a single-center experience. Dig Dis Sci. 2012 Mar;57(3):732-7. doi: 10.1007/s10620-011-1917-2. Epub 2011 Sep 30. PMID 21960285
- [Background] Na HK, Kim DH, Ahn JY, Lee JH, Jung KW, Choi KD, Song HJ, Lee GH, Jung HY. Clinical Outcomes following Endoscopic Treatment for Sporadic Nonampullary Duodenal Adenoma. Dig Dis. 2020;38(5):364-372. doi: 10.1159/000504249. Epub 2020 Jun 9. PMID 32516770
- [Background] Manner H, Enderle MD, Pech O, May A, Plum N, Riemann JF, Ell C, Eickhoff A. Second-generation argon plasma coagulation: two-center experience with 600 patients. J Gastroenterol Hepatol. 2008 Jun;23(6):872-8. doi: 10.1111/j.1440-1746.2008.05437.x. PMID 18565020
- [Background] Eickhoff A, Hartmann D, Eickhoff JC, Riemann JF, Enderle MD. Pain sensation and neuromuscular stimulation during argon plasma coagulation in gastrointestinal endoscopy. Surg Endosc. 2008 Jul;22(7):1701-7. doi: 10.1007/s00464-007-9700-3. Epub 2007 Dec 11. PMID 18071803
- [Background] Amoyel M, Belle A, Dhooge M, Ali EA, Hallit R, Prat F, Dohan A, Terris B, Chaussade S, Coriat R, Barret M. Endoscopic management of non-ampullary duodenal adenomas. Endosc Int Open. 2022 Jan 14;10(1):E96-E108. doi: 10.1055/a-1723-2847. eCollection 2022 Jan. PMID 35047339
- [Background] Kim GE, Siddiqui UD. Endoscopic Resection Techniques for Duodenal and Ampullary Adenomas. VideoGIE. 2023 Jul 22;8(8):330-335. doi: 10.1016/j.vgie.2023.05.006. eCollection 2023 Aug. PMID 37575136
- See also: German oncological guidelines for colorectal cancer — http://www.leitlinienprogramm-onkologie.de/leitlinien/kolorektales-karzinom/